CLINICAL TRIAL: NCT06395311
Title: The Impact of COPD on Psychological Well-being: A Cross-Sectional Study
Brief Title: Psychological Distress in Patients With COPD
Status: Completed | Type: Observational
Sponsor: Spitalul Clinic de Boli Infecțioase și Pneumoftiziologie Dr. Victor Babeș Timișoara (Other Government)
Responsible Party: Principal Investigator, Crisan Alexandru Florian, Principal Investigator, Spitalul Clinic de Boli Infecțioase și Pneumoftiziologie Dr. Victor Babeș Timișoara
Other Study IDs: 2045/11.03.2024
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: COPD; Quality of Life; Mental Health; Psychological Distress
Keywords: COPD; Quality of life; Anxiety and depression; Psychological distress
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Psychological Well-Being; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD subjects: Diagnosis of COPD established by a qualified healthcare professional (e.g., pulmonologist, general practitioner) based on:
  Post-bronchodilator spirometry demonstrating airflow obstruction (FEV1/FVC < 0.70) following GOLD (Global Initiative for Chronic Obstructive Lung Disease) guidelines.
  Age: 18 years or older. Adequate visual and/or auditory abilities to read and understand study materials/questionnaires or receive instructions verbally
  Interventions: Other: COPD psychological well-being assessment

INTERVENTIONS:
Other: COPD psychological well-being assessment — Patients will complete the following questionnaires: Hospital Anxiety and Depression Scale (HADS), COPD Assessment Test (CAT), State Shame and Guilt Scale (SSGS), Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE), Brief Fear of Negative Evaluation Scale (BFNE), Self-Compassion Scale Short Form (SCS-SF). Dyspnea will be evaluated with the mMRC scale, and functional capacity will be assessed with the six-minute walking test (6MWT).

SUMMARY:
Chronic obstructive pulmonary disease (COPD) can significantly impact a person's quality of life, not only physically but also mentally. This cross-sectional study aims to assess the psychological well-being of COPD patients by utilising specific questionnaires. These questionnaires will evaluate various aspects of mental health, including anxiety, depression, and potentially other relevant factors like self-compassion or fear of negative evaluation, self-efficacy, shame, and guilt. Additionally, the study will examine how these psychological factors relate to the severity of COPD symptoms, such as dyspnea and functional limitations. By understanding the psychological impact of COPD, this research hopes to emphasize the importance of medical education and mental health support in COPD management strategies.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) profoundly impacts both physical health and quality of life. Beyond the challenges of breathlessness and functional limitations, COPD patients often struggle with anxiety, depression, and other mental health difficulties at a much higher rate than the general population. This cross-sectional study seeks to understand the current state of psychological well-being in patients with COPD and explore how it relates to the severity of their condition. the study aims to assess the psychological well-being of COPD patients by utilizing specific questionnaires. These questionnaires will evaluate various aspects of mental health, including anxiety, depression, and potentially other relevant factors like self-compassion or fear of negative evaluation, self-efficacy, shame, and guilt. Additionally, the study will examine how these psychological factors relate to the severity of COPD symptoms, such as dyspnea and functional limitations. Investigators will use the following tests:

1. The Hospital Anxiety and Depression Scale (HADS) to identify and measure the severity of anxiety and depression symptoms.
2. The COPD Assessment Test (CAT) to measure the impact of COPD on a person's well-being.
3. The State Shame and Guilt Scale (SSGS) to measure a person's shame and guilt.
4. The Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE) to measure the patient's self-efficacy in managing their chronic respiratory disease.
5. The Brief Fear of Negative Evaluation Scale (BFNE) to assess an individual's anxiety around being judged or criticized by others.
6. The Self-Compassion Scale Short Form (SCS-SF) to measure key components of self-compassion.
7. The mMRC scale to evaluate the patient's level of breathlessness (dyspnea) in everyday life.
8. The six-minute walking test (6MWT) to measure how far a person can walk on a flat, hard surface in six minutes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD established by a qualified healthcare professional (e.g., pulmonologist, general practitioner) based on:
* Post-bronchodilator spirometry demonstrating airflow obstruction (FEV1/FVC < 0.70) following GOLD (Global Initiative for Chronic Obstructive Lung Disease) guidelines.
* Age: 40 years or older.
* Adequate visual and/or auditory abilities to read and understand study materials and questionnaires or receive instructions verbally if needed.

Exclusion Criteria:

* Other major respiratory illnesses: diagnosis of severe asthma, cystic fibrosis, lung cancer, or other significant respiratory diseases that could present with distinct psychological profiles.
* Acute COPD exacerbation: experiencing an acute exacerbation of COPD symptoms within the past four weeks.
* Unstable comorbid conditions: the presence of severe, uncontrolled medical conditions that could significantly affect cognitive function, well-being, or the ability to participate (e.g., unstable heart failure, end-stage renal disease, rapidly progressing malignancy).
* Severe mental disorders: current or recent diagnosis of a major psychiatric disorder that could significantly interfere with the interpretation of psychological measures or the ability to provide reliable responses (e.g., active schizophrenia, bipolar disorder, a major depressive episode).
* Problematic substance abuse: current problematic alcohol or illicit drug use (including opioids).
* Inability to provide informed consent: individuals lacking the cognitive capacity to understand the study and provide consent.
* Limited language proficiency: insufficient understanding of the language in which the study materials, including questionnaires, are administered.

Ages: 40 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with COPD post-bronchodilator spirometry demonstrating airflow obstruction (FEV1/FVC < 0.70) following GOLD (Global Initiative for Chronic Obstructive Lung Disease) guidelines.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression assessment | At inclusion
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment questionnaire used to identify and measure the severity of anxiety and depression symptoms. It has 14 questions, divided into seven questions assessing anxiety (HADS-A) and seven questions assessing depression (HADS-D). Each question has a 4-point response scale (0-3). Scores of 0-7: normal, scores of 8-10: suggestive of anxiety or depression, and scores of 11+ indicate probable presence of anxiety or depression.
Impact of COPD | At inclusion
  The COPD Assessment Test (CAT) is a questionnaire designed to measure the impact of COPD on a person's well-being. It consists of 8 simple questions. Each question has a 6-point scale (0-5) for the patient to rate their experience. Total scores range from 0 to 40. Higher scores indicate a greater negative impact of COPD on a person's life.
Shame and guilt assessment | At inclusion
  The State Shame and Guilt Scale (SSGS) is a self-report questionnaire that measures a person's shame and guilt. It has 15 questions in total, divided into three subscales: shame (5 questions), guilt (5 questions), and pride (5 questions), which measures the opposite of shame and guilt. Each item has a 5-point Likert scale ranging from 1 (not feeling in this way) to 5 (feeling this way very strongly). Higher scores on each subscale mean individuals experience those feelings more strongly in the moment.
Self-efficacy assessment | At inclusion
  The Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE) is a questionnaire designed to measure a patient's self-efficacy in managing their chronic respiratory disease, particularly within the context of pulmonary rehabilitation. It has 12 questions focused on managing breathlessness, staying physically active, and coping with emotional challenges due to respiratory disease. Patients rate their confidence on a scale of 1 to 10. Higher scores indicate greater self-efficacy.
Fear of negative evaluation assessment | At inclusion
  The Brief Fear of Negative Evaluation Scale (BFNE) is a psychological tool used to assess an individual's anxiety around being judged or criticized by others. It consists of 12 items. Statements capture different aspects of fear of negative evaluation. The scale uses a Likert scale response format (e.g., 1 = Not at all characteristic of me, 5 = Extremely characteristic of me). Scores are calculated by summing the responses to each item. Higher scores indicate a greater fear of negative evaluation.
Self-compassion assessment | At inclusion
  The Self-Compassion Scale Short Form (SCS-SF) is designed to measure key components of self-compassion. It consists of 12 items. Two items measure each of the six aspects of self-compassion: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. It uses a 5-point Likert scale (1 = almost never to 5 = almost always). A total self-compassion score is calculated. Higher scores indicate greater self-compassion.
Dyspnea assessment | At inclusion
  The mMRC scale is a simple questionnaire that grades a patient's level of breathlessness (dyspnea) in everyday life. It has five grades (0-4). The patient selects the statement that best aligns with their experience of breathlessness. Higher scores on the mMRC scale correlate to an increased level of disability for the patient due to breathlessness.
Aerobic capacity assessment | At inclusion
  The six-minute walking test (6MWT) measures how far a person can walk on a flat, hard surface in six minutes. It is used to assess aerobic capacity and functional endurance (how well the body can handle activity). The distance walked in 6 minutes is compared with predicted values based on age, gender, and height. A shorter walking distance indicates a lower level of functional exercise capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Crișan, PhD, Principal Investigator — Spitalul Clinic de Boli Infecțioase și Pneumoftiziologie Dr. Victor Babeș Timișoara
Locations (1):
- Spitalul de Boli Infectioase si Pneumoftiziologie Victor Babes, Timișoara, Timiș County, Romania